CLINICAL TRIAL: NCT04754594
Title: A PHASE 2/3, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLIND STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A SARS-COV-2 RNA VACCINE CANDIDATE (BNT162b2) AGAINST COVID-19 IN HEALTHY PREGNANT WOMEN 18 YEARS OF AGE AND OLDER
Brief Title: To Evaluate the Safety, Tolerability, and Immunogenicity of BNT162b2 Against COVID-19 in Healthy Pregnant Women 18 Years of Age and Older
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4591015; 2020-005444-35 (EudraCT Number)
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: SARS-CoV-2 Infection; COVID-19; Maternal Immunization
Keywords: SARS-CoV-2 Infection; COVID-19; Maternal Immunization
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BNT162b2 (Experimental): 2 doses
  Interventions: Biological: BNT162b2
- Placebo (Placebo Comparator): 2 doses
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT162b2 — Intramuscular Injection
  Arms: BNT162b2
Other: Placebo — Intramuscular Injection
  Arms: Placebo

SUMMARY:
Results will be submitted, however please note that data are not yet available for all serology outcome measures.

This will be a Phase 2/3, randomized, placebo-controlled, observer-blind study evaluating the safety, tolerability, and immunogenicity of 30 µg of BNT162b2 or placebo administered in 2 doses, 21 days apart, in approximately 350 healthy pregnant women 18 years of age or older vaccinated at 24 to 34 weeks' gestation. Participants will be randomized 1:1 to receive BNT162b2 or placebo (saline).

DETAILED DESCRIPTION:
The Phase 2 portion of the study will include approximately 200 pregnant women randomized 1:1 to receive BNT162b2 or placebo (saline) at 27 to 34 weeks' gestation. IRC review of safety data through 7 days after the second dose for all Phase 2 participants will be completed.

The Phase 3 portion of this study will assess the safety, tolerability, and immunogenicity of BNT162b2 among pregnant women enrolled at 24 to 34 weeks' gestation.

Maternal participants who originally received placebo will receive BNT162b2 at defined time points as part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women ≥18 years of age who are between 24 0/7 and 34 0/7 weeks' gestation on the day of planned vaccination, with an uncomplicated, singleton pregnancy, who are at no known increased risk for complications.
2. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Healthy participants who are determined by medical history, physical examination, and clinical judgment to be appropriate for inclusion in the study
4. Documented negative HIV antibody test (Phase 2 only), syphilis test, and HBV surface antigen test during this pregnancy and prior to randomization
5. Participant is willing to give informed consent for her infant to participate in the study
6. Capable of giving signed informed consent

Exclusion Criteria:

1. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
2. Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID 19.
3. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention or any related vaccine.
4. Participants with known or suspected immunodeficiency.
5. Bleeding diathesis or condition associated with prolonged bleeding that would in the opinion of the investigator contraindicate intramuscular injection.
6. Previous vaccination with any coronavirus vaccine.
7. Receipt of medications intended to prevent COVID 19.
8. Receipt of blood/plasma products or immunoglobulin, from 60 days before administration of study intervention, or planned receipt through delivery, with 1 exception, anti-D immunoglobulin (eg, RhoGAM), which can be given at any time.
9. Current alcohol abuse or illicit drug use.
10. Participants who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt through the postvaccination blood draw.
11. Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
12. Previous participation in other studies involving study intervention containing LNPs.
13. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
14. Participants whose unborn baby has been fathered by investigational site staff members directly involved in the conduct of the study or their family members, site staff members otherwise supervised by the investigator, or Pfizer employees directly involved in the conduct of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 726 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (87):
- United States (55):
  - Children's of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Women & Infant Center, Birmingham, Alabama
  - University of Alabama at Birmingham/Center for Women's Reproductive Health, Birmingham, Alabama
  - Velocity Clinical Research, Gulfport, Mobile, Alabama
  - Arrowhead Hospital, Glendale, Arizona
  - Abrazo West Campus Hospital, Goodyear, Arizona
  - St. Joseph Hospital, Phoenix, Arizona
  - MedPharmics, LLC, Phoenix, Arizona
  - Matrix Clinical Research., Huntington Park, California
  - Matrix Clinical Research, Huntington Park, California
  - Chemidox Clinical Trials Inc., Lancaster, California
  - East LA Doctors Hospital, Los Angeles, California
  - Matrix Clinical Research, Los Angeles, California
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Idaho Falls Pediatrics, Ammon, Idaho
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Idaho Falls Pediatrics, Idaho Falls, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - Mountain View Hospital, Idaho Falls, Idaho
  - Covenant Healthcare, Saginaw, Michigan
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Community Hospital of Anaconda, Anaconda, Montana
  - Boeson Research (BUT), Butte, Montana
  - SCL St. James Healthcare Hospital, Butte, Montana
  - Marcus Daly Memorial Hospital, Hamilton, Montana
  - Providence St. Patrick Hospital, Missoula, Montana
  - The Birth Center, Missoula, Montana
  - Boeson Research, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Community Physicians Group-Maternal Fetal Medicine, Missoula, Montana
  - St. Luke Community Healthcare Hospital, Ronan, Montana
  - Meridian Clinical Research, LLC, Hastings, Nebraska
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - OBGYN Associates of Erie, Erie, Pennsylvania
  - Central Erie Primary Care, Erie, Pennsylvania
  - Liberty Family Practice, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - St. David's Medical Center, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - Texas Health Harris Methodist Hospital Hurst-Euless-Bedford, Bedford, Texas
  - Ventavia Research Group LLC, Dallas, Texas
  - DHR Health Institute for Research and Development, Edinburg, Texas
  - 8th Avenue Obstetrics & Gynecology, Fort Worth, Texas
  - Baylor Scott & White All Saints Medical Center, Fort Worth, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Dr. Ruben Aleman & Associates, McAllen, Texas
  - Ventavia Research Group, LLC, Plano, Texas
  - Ventavia Research Group, LLC, Weatherford, Texas
  - Weatherford OBGYN, Weatherford, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - The Group for Women- MAWC, Norfolk, Virginia
  - Tidewater Physicians for Women- MAWC, Norfolk, Virginia
- Brazil (7):
  - Faculdade de Medicina da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - HMU SBC - Hospital Municipal Universitário de São Bernardo, São Bernardo do Campo, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo, São Paulo
  - Hospital Santa Casa de Misericordia de Sorocaba, Sorocaba, São Paulo
  - Clinica de Alergia Martti Antila S/S Ltda./ CMPC - Consultoria Medica e Pesquisa Clinica, Sorocaba, São Paulo
  - Unimed Sorocaba-Hospital Dr. Miguel Soeiro (HMS), Sorocaba, São Paulo
- South Africa (6):
  - WorthWhile Clinical Trials, Benoni, Gauteng
  - Wits Reproductive Health and HIV Institute (Wits RHI) Shandukani Research Centre, Johannesburg, Gauteng
  - Botho Ke Bontle Health Services, Pretoria, Gauteng
  - Vaccines and Infectious Diseases Analytics (VIDA), Soweto, Gauteng
  - Dr Tobias de Villiers, Cape Town, Western Cape
  - Tiervlei Trial Centre CC, Cape Town, Western Cape
- Spain (12):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Hospital de Antequera, Antequera, Malaga
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Clinica Diagonal, Barcelona
  - Hospital Madrid Puerta del Sur Mostoles, Móstoles
  - Instituto Hispalense de Pediatria- IHP1, Seville
  - Hospital Materno-Infantil Quirón, Seville
  - Servicio de Ginecología del Hospital Quirón Salud Sagrado Corazón, Seville
- United Kingdom (7):
  - Hampshire Research Hub, Royal South Hants Hospital, Southampton, Hampshire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Medway NHS Foundation Trust, Gillingham, KENT
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University College London Hospitals, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nana M, Hodson K, Lucas N, Camporota L, Knight M, Nelson-Piercy C. Diagnosis and management of covid-19 in pregnancy. BMJ. 2022 Apr 26;377:e069739. doi: 10.1136/bmj-2021-069739. PMID 35473709
- [Derived] Mohapatra S, Ananda P, Tripathy S. Pharmacological consideration of COVID-19 infection and vaccines in pregnancy. J Chin Med Assoc. 2022 May 1;85(5):537-542. doi: 10.1097/JCMA.0000000000000712. Epub 2022 May 2. PMID 35316227
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 2 periods-Blinded Period (from Day 1 to 1 month post-delivery) and Unblinded Period (1 to 6 Months Post-Delivery for those maternal participants who initially received BNT162b2 and from first dose of BNT162b2 to 1 month after second dose of BNT162b2 for those maternal participants who initially received placebo).
Pre-assignment Details: A total of 726 participants were enrolled in this study. 391 were maternal participants who signed informed consent form and were enrolled out of which 41 were screen failures and 2 participants were not randomized. Eventually 348 maternal participants were randomized to receive treatment. 335 were infants born to maternal participants.
Groups:
- Maternal Participants: BNT162b2 30 mcg: Maternal participants received two doses of BNT162b2 30 micrograms (mcg) as an intramuscular injection separated by 21 days during their 24 to 34 weeks gestation in the blinded phase. Participants were followed-up until 6 months post-delivery.
- Maternal Participants: Placebo Then BNT162b2 30 mcg: Maternal participants received two doses of placebo as an intramuscular injection separated by 21 days during their 24 to 34 weeks gestation in the blinded phase. After unblinding at 1 month post-delivery, participants were administered 2 doses of BNT162b2 vaccine as an intramuscular injection separated by 21 days. Participants were followed-up until 1 month after last dose of vaccination.
- Infant Participants: BNT162b2 30 mcg: Infant participants who were born to maternal participants vaccinated with BNT162b2 30 mcg during pregnancy were included. Infant participants were followed up to 6 months of age.
- Infant Participants: Placebo: Infant participants who were born to maternal participants vaccinated with placebo during pregnancy were included. Infant participants were followed up to 6 months of age.
Period: Blinded Period
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo Then BNT162b2 30 mcg | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo
Started | 174 | 174 | 0 | 0
Vaccination 1 | 173 | 173 | 0 | 0
Vaccination 2 | 170 | 170 | 0 | 0
Completed | 161 | 159 | 0 | 0
Not Completed | 13 | 15 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 9 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Unblinded before 1-month postdelivery visit | 6 | 3 | 0 | 0
Period: Unblinded Period
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo Then BNT162b2 30 mcg | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo
Started | 167 (6 participants unblinded before 1-month post delivery are also included.) | 162 (3 participants unblinded before 1-month post delivery are also included.) | 0 | 0
Vaccination 3 | 0 | 152 | 0 | 0
Vaccination 4 | 0 | 148 | 0 | 0
Completed | 151 | 147 | 0 | 0
Not Completed | 16 | 15 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 8 | 0 | 0
Not completed — Lost to Follow-up | 5 | 3 | 0 | 0
Not completed — Protocol Violation | 2 | 4 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0
Period: Infant Participants
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo Then BNT162b2 30 mcg | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo
Started | 0 | 0 | 167 | 168
Completed | 0 | 0 | 152 | 139
Not Completed | 0 | 0 | 15 | 29
Not completed — Withdrawal by Subject | 0 | 0 | 9 | 17
Not completed — Lost to Follow-up | 0 | 0 | 4 | 10
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: For maternal participants, safety population included all randomized participants who received at least 1 dose of the study intervention. For infant participants, safety population included all infant participants born to maternal participants who received at least 1 dose of the study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo Then BNT162b2 30 mcg | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo | Total
Number analyzed (Participants) | 173 | 173 | 167 | 168 | 681
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 18 years | 0 | 0 | 167 | 168 | 335
  Greater than or equal to (>=) 18 and <= 45 years | 173 | 173 | 0 | 0 | 346
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 173 | 85 | 73 | 504
  Male | 0 | 0 | 82 | 95 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 63 | 65 | 60 | 258
  Not Hispanic or Latino | 103 | 110 | 98 | 104 | 415
  Unknown or Not Reported | 0 | 0 | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 2 | 5
  Asian | 5 | 9 | 3 | 7 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 47 | 43 | 40 | 40 | 170
  White | 117 | 118 | 115 | 104 | 454
  More than one race | 1 | 0 | 0 | 6 | 7
  Unknown or Not Reported | 2 | 1 | 8 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Maternal Participants Reporting Local Reactions Within 7 Days After Dose 1
Description: Pain at injection site, redness & swelling were recorded by participants in an electronic diary (e-diary). Redness & swelling were measured & recorded in measuring devise units (range 1 to 21) then converted to cm. 1 measuring device unit = 0.5 cm & graded as mild: > 2.0 to 5.0 cm, moderate: > 5.0 to 10.0 cm, severe: > 10.0 cm, grade 4 (potentially life threatening): necrosis or exfoliative dermatitis (redness) & necrosis (swelling). Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity & grade 4 (potentially life threatening): emergency room visit or hospitalization for severe pain. Grade 4 reactions were classified by the investigator or medically qualified person. Reactions reported as adverse events in the case report form within 7 days after the study vaccination were also included in the analysis. Exact 2-sided 95% confidence interval (CI) was based on Clopper & Pearson method.
Time Frame: From Day 1 to Day 7 after dose 1
Population: For maternal participants, safety population included all randomized participants who received at least 1 dose of the study intervention. Here, "Overall Number of Participants Analyzed" (N) signifies participants evaluable for this outcome measure. Human immunodeficiency virus (HIV) positive participants were excluded from analysis as pre-specified in the statistical analysis plan (SAP).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Maternal Participants: Placebo: Maternal participants received two doses of placebo as an intramuscular injection separated by 21 days during their 24 to 34 weeks gestation in the blinded phase.
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 161 | 163
Percentage of participants
  Redness: Mild | 2.5 [0.7 to 6.2] | 0.6 [0.0 to 3.4]
  Redness: Moderate | 0.6 [0.0 to 3.4] | 0 [0.0 to 2.2]
  Redness: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Redness: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Swelling: Mild | 4.3 [1.8 to 8.8] | 0 [0.0 to 2.2]
  Swelling: Moderate | 0.6 [0.0 to 3.4] | 0 [0.0 to 2.2]
  Swelling: Severe | 0.6 [0.0 to 3.4] | 0 [0.0 to 2.2]
  Swelling: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Pain at the injection site: Mild | 59.0 [51.0 to 66.7] | 9.8 [5.7 to 15.5]
  Pain at the injection site: Moderate | 23.6 [17.3 to 30.9] | 0 [0.0 to 2.2]
  Pain at the injection site: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Pain at the injection site: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]

2. Primary Outcome: Percentage of Maternal Participants Reporting Local Reactions Within 7 Days After Dose 2
Description: Pain at injection site, redness & swelling were recorded by participants in an e-diary. Redness & swelling were measured & recorded in measuring devise units (range 1 to 21) then converted to cm. 1 measuring device unit = 0.5 cm & graded as mild: > 2.0 to 5.0 cm, moderate: > 5.0 to 10.0 cm, severe: > 10.0 cm, grade 4 (potentially life threatening): necrosis or exfoliative dermatitis (redness) & necrosis (swelling). Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity & grade 4 (potentially life threatening): emergency room visit or hospitalization for severe pain. Grade 4 reactions were classified by the investigator or medically qualified person. Reactions reported as adverse events (AEs) in the case report form (CRF) within 7 days after the study vaccination were also included in the analysis. Exact 2-sided 95% CI was based on the Clopper & Pearson method.
Time Frame: From Day 1 to Day 7 after dose 2
Population: For maternal participants, safety population included all randomized participants who received at least 1 dose of the study intervention. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. HIV positive participants were excluded from analysis as pre-specified in the SAP.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 148 | 146
Percentage of participants
  Redness: Mild | 3.4 [1.1 to 7.7] | 0 [0.0 to 2.5]
  Redness: Moderate | 2.0 [0.4 to 5.8] | 0 [0.0 to 2.5]
  Redness: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Redness: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Swelling: Mild | 4.1 [1.5 to 8.6] | 0.7 [0.0 to 3.8]
  Swelling: Moderate | 2.7 [0.7 to 6.8] | 0 [0.0 to 2.5]
  Swelling: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Swelling: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Pain at the injection site: Mild | 54.7 [46.3 to 62.9] | 12.3 [7.5 to 18.8]
  Pain at the injection site: Moderate | 19.6 [13.5 to 26.9] | 4.1 [1.5 to 8.7]
  Pain at the injection site: Severe | 0.7 [0.0 to 3.7] | 0 [0.0 to 2.5]
  Pain at the injection site: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]

3. Primary Outcome: Percentage of Maternal Participants Reporting Systemic Events Within 7 Days After Dose 1
Description: Systemic events were recorded by participants in an e-diary. Fever was oral temperature >= 38 degree Celsius (°C) & categorized as >=38.0 to 38.4 °C, >38.4 to 38.9 °C, >38.9 to 40.0 °C & >40.0 °C. Fatigue, headache, chills, new or worsened muscle pain & new or worsened joint pain were graded mild: did not interfere with activity, moderate: some interference with activity & severe: prevented daily routine activity. Vomiting was graded mild: 1 to 2 times in 24 hours (h), moderate: >2 times in 24h & severe: required intravenous hydration. Diarrhea was graded mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h & severe: 6 or more loose stools in 24h. For all systemic events except fever, Grade 4= emergency room visit or hospitalization. Grade 4 events were classified by the investigator/medically qualified person. Systemic events reported as AEs in the CRF within 7 days after vaccination were also included in analysis. Exact 95% CI was based on Clopper & Pearson method.
Time Frame: From Day 1 to Day 7 after dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 161 | 163
Percentage of participants
  Fever: >=38.0 to 38.4 deg C (100.4 to 101.1 deg Fahrenheit [F]) | 0.6 [0.0 to 3.4] | 1.2 [0.1 to 4.4]
  Fever: >38.4 to 38.9 deg C (101.2 to 102.0 deg F) | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Fever: >38.9 to 40.0 deg C (102.1 to 104.0 deg F) | 0.6 [0.0 to 3.4] | 0.6 [0.0 to 3.4]
  Fever: >40 deg C (>104.0 deg F) | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Fatigue/tiredness: Mild | 26.1 [19.5 to 33.6] | 20.9 [14.9 to 27.9]
  Fatigue/tiredness: Moderate | 23.0 [16.7 to 30.3] | 21.5 [15.4 to 28.6]
  Fatigue/tiredness: Severe | 0.6 [0.0 to 3.4] | 0.6 [0.0 to 3.4]
  Fatigue/tiredness: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Headache: Mild | 20.5 [14.5 to 27.6] | 22.1 [16.0 to 29.2]
  Headache: Moderate | 11.8 [7.3 to 17.8] | 12.9 [8.2 to 19.0]
  Headache: Severe | 1.9 [0.4 to 5.3] | 0.6 [0.0 to 3.4]
  Headache: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Chills: Mild | 5.0 [2.2 to 9.6] | 5.5 [2.6 to 10.2]
  Chills: Moderate | 1.9 [0.4 to 5.3] | 0 [0.0 to 2.2]
  Chills: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Chills: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Vomiting: Mild | 5.0 [2.2 to 9.6] | 6.1 [3.0 to 11.0]
  Vomiting: Moderate | 0 [0.0 to 2.3] | 3.1 [1.0 to 7.0]
  Vomiting: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Vomiting: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Diarrhea: Mild | 11.2 [6.8 to 17.1] | 7.4 [3.9 to 12.5]
  Diarrhea: Moderate | 0.6 [0.0 to 3.4] | 1.2 [0.1 to 4.4]
  Diarrhea: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  Diarrhea: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  New or worsened muscle pain: Mild | 6.8 [3.5 to 11.9] | 6.1 [3.0 to 11.0]
  New or worsened muscle pain: Moderate | 5.6 [2.6 to 10.3] | 5.5 [2.6 to 10.2]
  New or worsened muscle pain: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  New or worsened joint pain: Mild | 1.2 [0.2 to 4.4] | 2.5 [0.7 to 6.2]
  New or worsened joint pain: Moderate | 1.9 [0.4 to 5.3] | 2.5 [0.7 to 6.2]
  New or worsened joint pain: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 2.2]

4. Primary Outcome: Percentage of Maternal Participants Reporting Systemic Events Within 7 Days After Dose 2
Description: Systemic events were recorded by participants in an e-diary. Fever was oral temperature >= 38 °C & categorized as >=38.0 to 38.4 °C, >38.4 to 38.9 °C, >38.9 to 40.0 °C & >40.0 °C. Fatigue, headache, chills, new or worsened muscle pain & new or worsened joint pain were graded mild: did not interfere with activity, moderate: some interference with activity & severe: prevented daily routine activity. Vomiting was graded mild: 1 to 2 times in 24 h, moderate: >2 times in 24 h & severe: required intravenous hydration. Diarrhea was graded mild: 2 to 3 loose stools in 24 h, moderate: 4 to 5 loose stools in 24 h & severe: 6 or more loose stools in 24 h. For all systemic events except fever, Grade 4= emergency room visit or hospitalization. Grade 4 events were classified by the investigator/medically qualified person. Systemic events reported as AEs in the CRF within 7 days after vaccination were also included in analysis. Exact 95% CI was based on Clopper & Pearson method.
Time Frame: From Day 1 to Day 7 after dose 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 148 | 146
Percentage of participants
  Fever: >=38.0 to 38.4 deg C (100.4 to 101.1 deg F) | 1.4 [0.2 to 4.8] | 0.7 [0.0 to 3.8]
  Fever: >38.4 to 38.9 deg C (101.2 to 102.0 deg F) | 0.7 [0.0 to 3.7] | 0 [0.0 to 2.5]
  Fever: >38.9 to 40.0 deg C (102.1 to 104.0 deg F) | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Fever: >40 deg C (>104.0 deg F) | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Fatigue/tiredness: Mild | 15.5 [10.1 to 22.4] | 15.8 [10.3 to 22.7]
  Fatigue/tiredness: Moderate | 32.4 [25.0 to 40.6] | 18.5 [12.6 to 25.8]
  Fatigue/tiredness: Severe | 2.0 [0.4 to 5.8] | 0 [0.0 to 2.5]
  Fatigue/tiredness: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Headache: Mild | 25.0 [18.3 to 32.8] | 13.7 [8.6 to 20.4]
  Headache: Moderate | 14.9 [9.6 to 21.6] | 10.3 [5.9 to 16.4]
  Headache: Severe | 1.4 [0.2 to 4.8] | 0 [0.0 to 2.5]
  Headache: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Chills: Mild | 4.7 [1.9 to 9.5] | 0.7 [0.0 to 3.8]
  Chills: Moderate | 7.4 [3.8 to 12.9] | 0 [0.0 to 2.5]
  Chills: Severe | 0.7 [0.0 to 3.7] | 0 [0.0 to 2.5]
  Chills: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Vomiting: Mild | 8.8 [4.8 to 14.6] | 2.1 [0.4 to 5.9]
  Vomiting: Moderate | 0 [0.0 to 2.5] | 1.4 [0.2 to 4.9]
  Vomiting: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Vomiting: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Diarrhea: Mild | 6.1 [2.8 to 11.2] | 4.1 [1.5 to 8.7]
  Diarrhea: Moderate | 0 [0.0 to 2.5] | 1.4 [0.2 to 4.9]
  Diarrhea: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Diarrhea: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  New or worsened muscle pain: Mild | 13.5 [8.5 to 20.1] | 4.8 [1.9 to 9.6]
  New or worsened muscle pain: Moderate | 12.8 [7.9 to 19.3] | 2.1 [0.4 to 5.9]
  New or worsened muscle pain: Severe | 0.7 [0.0 to 3.7] | 0 [0.0 to 2.5]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  New or worsened joint pain: Mild | 7.4 [3.8 to 12.9] | 4.8 [1.9 to 9.6]
  New or worsened joint pain: Moderate | 6.1 [2.8 to 11.2] | 1.4 [0.2 to 4.9]
  New or worsened joint pain: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]

5. Primary Outcome: Percentage of Maternal Participants With Adverse Events (AEs) From Dose 1 Through 1 Month After Dose 2 - Blinded Follow-up Period
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From dose 1 on Day 1 through 1 month after dose 2 (approximately 2 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 161 | 163
Percentage of participants | 23.6 [17.3 to 30.9] | 22.7 [16.5 to 29.9]

6. Primary Outcome: Percentage of Maternal Participants Reporting Serious Adverse Events (SAEs) From Dose 1 Through 1 Month After Delivery - Blinded Follow-up Period
Description: An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening; resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required inpatient hospitalization or prolongation of existing hospitalization. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: From dose 1 on Day 1 through 1 month after delivery (up to 22 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 161 | 163
Percentage of participants | 13.0 [8.3 to 19.2] | 14.1 [9.2 to 20.4]

7. Primary Outcome: Geometric Mean Ratio (GMR) of the SARS-CoV-2 Neutralizing Titers in Pregnant Women to Those in Nonpregnant Women From Study C4591001 (NCT04368728) for Evaluable Immunogenicity Population Without Evidence of Prior SARS-CoV-2 Infection
Description: GMR of SARS-CoV-2 neutralizing titers in pregnant women to those in nonpregnant women from study C4591001 (NCT04368728) for evaluable immunogenicity population without evidence of prior SARS-CoV-2 infection up to 1 month after Dose 2 was reported in this outcome measure. Geometric mean titer (GMT) and 2-sided 95% CIs were calculated by exponentiating mean logarithm of titers and corresponding CIs (based on student t distribution) and was reported in descriptive section. GMR was reported in statistical analysis section of this outcome measure. Evaluable immunogenicity population included all participants who were eligible and randomized, received 2 doses of vaccine to which they were randomized, with Dose 2 received within predefined window (19-42 days, inclusive, after Dose 1); had at least 1 valid immunogenicity result within an appropriate window 1 month after Dose 2 (28-42 days, inclusive, after Dose 2); and had no other important protocol deviations as determined by the clinician.
Time Frame: 1 Month after Dose 2
Population: Evaluable immunogenicity population without evidence of SARS-CoV2 infection up to 1 month after Dose 2 was analyzed. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. HIV positive participants were excluded from analysis as pre-specified in the SAP.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Maternal Participants: BNT162b2 30 mcg: Maternal participants received two doses of BNT162b2 30 micrograms (mcg) as an intramuscular injection separated by 21 days.
- Non-Pregnant Participants: Study C4591001: Non-pregnant participants who received two doses of BNT162b2 30 mcg as an intramuscular injection separated by 21 days in study C4591001 (NCT04368728).
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Non-Pregnant Participants: Study C4591001
Number analyzed (Participants) | 58 | 107
Titer | 1109.2 [849.2 to 1448.9] | 1663.7 [1411.5 to 1960.8]
Statistical Analysis 1: Comparison: Maternal Participants: BNT162b2 30 mcg vs Non-Pregnant Participants: Study C4591001; GMRs and 2-sided 95% CIs was calculated by exponentiating the mean difference of the logarithms of the assay and the corresponding CIs; Test type: Other; Geometric mean ratio = 0.67, 95% CI 2-sided [0.50 to 0.90]

8. Primary Outcome: GMR of SARS-CoV-2 Neutralizing Titers in Pregnant Women to Those in Nonpregnant Women From Study C4591001 (NCT04368728) for Evaluable Immunogenicity Population With and Without Evidence of Prior SARS-CoV-2 Infection
Description: GMR of SARS-CoV-2 neutralizing titers in pregnant women to those in nonpregnant women from study C4591001 (NCT04368728) for evaluable immunogenicity population with and without evidence of prior SARS-CoV-2 infection was reported in this outcome measure. GMT and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the student t distribution) and was reported in the descriptive section. GMR was reported in the statistical analysis section. Evaluable immunogenicity population included all participants who were eligible and randomized, received 2 doses of the vaccine to which they were randomized, with Dose 2 received within the predefined window (19-42 days, inclusive, after Dose 1); had at least 1 valid immunogenicity result within an appropriate window 1 month after Dose 2 (28-42 days, inclusive, after Dose 2); and had no other important protocol deviations as determined by the clinician.
Time Frame: 1 Month after Dose 2
Population: Evaluable immunogenicity population was analyzed. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. HIV positive participants were excluded from analysis as pre-specified in the SAP.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Non-Pregnant Participants: Study C4591001
Number analyzed (Participants) | 100 | 114
Titer | 2198.7 [1618.5 to 2987.0] | 1732.0 [1469.4 to 2041.5]
Statistical Analysis 1: Comparison: Maternal Participants: BNT162b2 30 mcg vs Non-Pregnant Participants: Study C4591001; [analysis description as in outcome 7, analysis 1]; Test type: Other; Geometric mean ratio = 1.27, 95% CI 2-sided [0.91 to 1.77]
Statistical Analysis 2: Comparison: Maternal Participants: BNT162b2 30 mcg vs Non-Pregnant Participants: Study C4591001; [analysis description as in outcome 7, analysis 1]; Test type: Other; Geometric mean ratio = 0.95, 95% CI 2-sided [0.69 to 1.30]

9. Secondary Outcome: COVID-19 Incidence Per 100 Person-Years of Blinded Follow up in Evaluable Maternal Participants Without Evidence of Prior SARS-CoV-2 Infection
Description: COVID-19 incidence per 100 person-years of blinded follow-up in evaluable maternal participants without evidence of prior SARS-CoV-2 infection prior to 7 days after receipt of Dose 2 was reported in this outcome measure.
Time Frame: From 7 days after Dose 2 up to 1 month after delivery (Surveillance time [100 person-year]: BNT162b2- 0.155, Placebo- 0.149)
Population: Evaluable efficacy population included all eligible randomized participants who received all vaccinations as randomized, with Dose 2 received within predefined window (within 19-42 days after Dose 1) and had no other important protocol deviations as determined by clinician on or before 7 days after Dose 2. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. HIV positive participants were excluded from analysis as pre-specified in SAP.
Measure: Number; unit: Events per 100 person-years
Groups:
- Maternal Participants: BNT162b2 30 mcg: Maternal participants received two doses of BNT162b2 30 micrograms (mcg) as an intramuscular injection separated by 21 days during their 24 to 34 weeks gestation in the blinded phase.
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 86 | 89
Events per 100 person-years | 12.903 | 13.423
Statistical Analysis 1: Comparison: Maternal Participants: BNT162b2 30 mcg vs Maternal Participants: Placebo; Test type: Other — Vaccine efficacy was estimated by 100*(1 - illness rate ratio [IRR]), where IRR=calculated ratio of confirmed COVID-19 illness per 1000 person-years of blinded follow-up in the active vaccine group to the corresponding illness rate in the placebo group; Vaccine efficacy = 3.8, 95% CI 2-sided [-1227.8 to 93.0]

10. Secondary Outcome: COVID-19 Incidence Per 100 Person-Years of Blinded Follow up in Evaluable Maternal Participants With or Without Evidence of Prior SARS-CoV-2 Infection
Description: COVID-19 incidence per 100 person-years of blinded follow-up in evaluable maternal participants with or without evidence of prior SARS-CoV-2 infection was reported in this outcome measure.
Time Frame: From 7 days after Dose 2 up to 1 month after delivery (Surveillance time [100 person-year]: BNT162b2- 0.270, Placebo- 0.263)
Population: as for outcome 9
Measure: Number; unit: Events per 100 person-years
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 145 | 149
Events per 100 person-years | 7.407 | 11.407
Statistical Analysis 1: Comparison: Maternal Participants: BNT162b2 30 mcg vs Maternal Participants: Placebo; Test type: Other — Vaccine efficacy was estimated by 100*(1 - IRR), where IRR=calculated ratio of confirmed COVID-19 illness per 1000 person-years of blinded follow-up in the active vaccine group to the corresponding illness rate in the placebo group; Vaccine efficacy = 35.1, 95% CI 2-sided [-466.5 to 94.6]

11. Secondary Outcome: Incidence of Asymptomatic Infection of SARS-CoV-2 Through 1 Month After Delivery in Evaluable Maternal Participants Without Evidence of Prior SARS-CoV-2 Infection
Description: Incidence of asymptomatic infection of SARS-CoV-2 through 1 month after delivery in evaluable maternal participants without evidence of prior SARS-CoV-2 infection prior to the first post-dose 2 N-binding test was reported in this outcome measure.
Time Frame: Up to 1 month after delivery (Surveillance time [100 person-year]: BNT162b2- 0.099, Placebo- 0.147)
Population: as for outcome 9
Measure: Number; unit: Events per 100 person-years
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 84 | 89
Events per 100 person-years | 40.404 | 68.027
Statistical Analysis 1: Comparison: Maternal Participants: BNT162b2 30 mcg vs Maternal Participants: Placebo; Test type: Other — [test comment as in outcome 10, analysis 1]; Vaccine efficacy = 40.9, 95% CI 2-sided [-104.9 to 86.5]

12. Secondary Outcome: Geometric Mean Concentration (GMCs) of Full-Length S-Binding Immunoglobulin G (IgG) Levels in Evaluable Maternal Participants
Description: GMCs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. GMCs of full-length S-binding IgG levels in evaluable maternal participants at baseline, 2 weeks after Dose 2, 1 month after Dose 2, at delivery, and 6 months after delivery was reported in this outcome measure. Evaluable immunogenicity population included all participants who were eligible and randomized, received 2 doses of the vaccine to which they were randomized, with Dose 2 received within the predefined window (19-42 days, inclusive, after Dose 1); had at least 1 valid immunogenicity result within an appropriate window 1 month after Dose 2 (28-42 days, inclusive, after Dose 2); and had no other important protocol deviations as determined by the clinician.
Time Frame: Baseline (before Dose 1), 2 weeks after Dose 2, 1 month after Dose 2, at delivery, and 6 months after delivery
Population: Evaluable immunogenicity population was analyzed. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows. HIV positive participants were excluded from analysis as pre-specified in the SAP.
Measure: Geometric Mean (95% Confidence Interval); unit: Units/milliliter (U/mL)
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 65 | 59
Units/milliliter (U/mL)
  Before Dose 1 | 2.4 [1.6 to 3.7] | 2.0 [1.4 to 2.8]
  2 weeks after Dose 2: number analyzed (Participants) | 41 | 35
  2 weeks after Dose 2 | 7802.0 [6273.3 to 9703.2] | 1.8 [1.1 to 3.1]
  1 month after Dose 2: number analyzed (Participants) | 36 | 31
  1 month after Dose 2 | 4281.0 [3234.7 to 5665.7] | 1.8 [1.1 to 2.9]
  At delivery: number analyzed (Participants) | 39 | 29
  At delivery | 2747.6 [2144.7 to 3520.0] | 1.7 [1.0 to 3.0]
  6 months after delivery: number analyzed (Participants) | 20 | 0
  6 months after delivery | 1639.4 [780.1 to 3445.4] |

13. Secondary Outcome: Geometric Mean Titer (GMTs) of SARS-CoV-2 Neutralizing Titers in Evaluable Maternal Participants
Description: GMTs, and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. GMTs of SARS-CoV-2 neutralizing titers in evaluable maternal participants at baseline, 2 weeks after Dose 2, 1 month after Dose 2, at delivery, and 6 months after delivery was reported in this outcome measure. Evaluable immunogenicity population included all participants who were eligible and randomized, received 2 doses of the vaccine to which they were randomized, with Dose 2 received within the predefined window (19-42 days, inclusive, after Dose 1); had at least 1 valid immunogenicity result within an appropriate window 1 month after Dose 2 (28-42 days, inclusive, after Dose 2); and had no other important protocol deviations as determined by the clinician.
Time Frame: Baseline (before Dose 1), 2 weeks after Dose 2, 1 month after Dose 2, at delivery, and 6 months after delivery
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 65 | 59
Titer
  Before Dose 1 | 47.6 [41.6 to 54.4] | 43.5 [43.5 to 43.5]
  2 weeks after Dose 2: number analyzed (Participants) | 41 | 35
  2 weeks after Dose 2 | 1991.8 [1456.3 to 2724.1] | 45.0 [42.0 to 48.3]
  1 month after Dose 2: number analyzed (Participants) | 36 | 31
  1 month after Dose 2 | 1212.6 [855.2 to 1719.4] | 43.5 [43.5 to 43.5]
  At delivery: number analyzed (Participants) | 39 | 29
  At delivery | 695.7 [500.6 to 966.8] | 43.5 [43.5 to 43.5]
  6 months after delivery: number analyzed (Participants) | 20 | 0
  6 months after delivery | 465.4 [168.6 to 1284.5] |

14. Secondary Outcome: Geometric Mean Fold Rise (GMFR) From Before Vaccination to Each Subsequent Time Point After Vaccination for Full-Length S-Binding IgG Levels in Evaluable Maternal Participants
Description: GMFRs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. GMFR from before vaccination to each subsequent time point after vaccination for full-length S-binding IgG levels in evaluable maternal participants at 2 weeks after Dose 2, 1 month after Dose 2, at delivery, and 6 months after delivery was reported in this outcome measure. Evaluable immunogenicity population included all participants who were eligible and randomized, received 2 doses of the vaccine to which they were randomized, with Dose 2 received within the predefined window (19-42 days, inclusive, after Dose 1); had at least 1 valid immunogenicity result within an appropriate window 1 month after Dose 2 (28-42 days, inclusive, after Dose 2); and had no other important protocol deviations as determined by the clinician.
Time Frame: From before dose 1 up to 2 weeks after Dose 2, 1 month after Dose 2, at delivery, and 6 months after delivery
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 58 | 54
Fold rise
  2 weeks after Dose 2 | 3618.7 [2489.1 to 5260.7] | 0.9 [0.8 to 1.1]
  1 month after Dose 2: number analyzed (Participants) | 50 | 49
  1 month after Dose 2 | 2276.4 [1545.5 to 3352.9] | 0.9 [0.8 to 1.1]
  At delivery: number analyzed (Participants) | 55 | 47
  At delivery | 1377.6 [948.6 to 2000.5] | 0.8 [0.6 to 1.0]
  6 months after delivery: number analyzed (Participants) | 26 | 0
  6 months after delivery | 650.3 [279.3 to 1514.3] |

15. Secondary Outcome: Geometric Mean Fold Rise (GMFR) From Before Vaccination to Each Subsequent Time Point After Vaccination for SARS-CoV-2 Neutralizing Titers in Evaluable Maternal Participants
Description: GMFRs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. GMFR from before vaccination to each subsequent time point after vaccination for SARS-CoV-2 neutralizing titers in evaluable maternal participants at 2 weeks after Dose 2, 1 month after Dose 2, at delivery, and 6 months after delivery was reported in this outcome measure. Evaluable immunogenicity population included all participants who were eligible and randomized, received 2 doses of the vaccine to which they were randomized, with Dose 2 received within the predefined window (19-42 days, inclusive, after Dose 1); had at least 1 valid immunogenicity result within an appropriate window 1 month after Dose 2 (28-42 days, inclusive, after Dose 2); and had no other important protocol deviations as determined by the clinician.
Time Frame: From before dose 1 up to 2 weeks after Dose 2, 1 month after Dose 2, at delivery, and 6 months after delivery
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Maternal Participants: BNT162b2 30 mcg | Maternal Participants: Placebo
Number analyzed (Participants) | 58 | 54
Fold rise
  2 weeks after Dose 2 | 43.7 [33.9 to 56.4] | 1.0 [1.0 to 1.1]
  1 month after Dose 2: number analyzed (Participants) | 50 | 49
  1 month after Dose 2 | 25.3 [18.9 to 33.9] | 1.0 [1.0 to 1.0]
  At delivery: number analyzed (Participants) | 55 | 47
  At delivery | 15.6 [12.1 to 20.1] | 1.0 [1.0 to 1.0]
  6 months after delivery: number analyzed (Participants) | 26 | 0
  6 months after delivery | 11.3 [5.0 to 25.4] |

16. Secondary Outcome: Percentage of Infant Participants Reporting Specific Birth Outcomes
Description: Percentage of infant participants reporting specific birth outcomes (normal, congenital malformation/anomaly, other neonatal problems) were reported in this outcome measure.
Time Frame: At birth
Population: Safety population for infant participants included all infant participants born to maternal participants who received at least 1 dose of the study intervention. As this outcome measure was measured at birth, HIV positive infant participants were included in this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo
Number analyzed (Participants) | 167 | 168
Percentage of participants
  Normal | 91.6 [86.3 to 95.3] | 89.3 [83.6 to 93.5]
  Congenital malformation/anomaly | 6.0 [2.9 to 10.7] | 3.6 [1.3 to 7.6]
  Other neonatal problem | 1.8 [0.4 to 5.2] | 6.5 [3.3 to 11.4]

17. Secondary Outcome: Percentage of Infant Participants Reporting Adverse Events From Birth Through 1 Month of Age
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: From birth through 1 month of age
Population: Safety population for infant participants included all infant participants born to maternal participants who received at least 1 dose of the study intervention. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. HIV positive participants were excluded from analysis as pre-specified in the SAP.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo
Number analyzed (Participants) | 156 | 159
Percentage of participants | 35.3 [27.8 to 43.3] | 37.1 [29.6 to 45.1]

18. Secondary Outcome: Percentage of Infant Participants Reporting Serious Adverse Events (SAE) From Birth Through 6 Months of Age
Description: as for outcome 6
Time Frame: From birth through 6 months of age
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo
Number analyzed (Participants) | 156 | 159
Percentage of participants | 13.5 [8.5 to 19.8] | 15.1 [9.9 to 21.6]

19. Secondary Outcome: Percentage of Infant Participants Reporting Adverse Event of Special Interest (AESI) From Birth Through 6 Months of Age
Description: Percentage of infant participants who reported AESI including major congenital anomalies and developmental delay from birth through 6 months of age were reported in this outcome measure. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: From birth through 6 months of age
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo
Number analyzed (Participants) | 156 | 159
Percentage of participants | 5.1 [2.2 to 9.9] | 1.3 [0.2 to 4.5]

20. Secondary Outcome: GMCs of Full-Length S-Binding IgG Levels at Birth and 6 Months of Age in Infant Participants Born to Evaluable Maternal Participants
Description: GMCs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. GMCs of full-length S-binding IgG levels at birth and 6 months of age in infant participants born to evaluable maternal participants was reported in this outcome measure.
Time Frame: At birth and 6 months of age
Population: All infant participants born to evaluable immunogenicity maternal participants and had no important protocol deviations as determined by the clinician. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows. HIV positive participants were excluded from analysis as pre-specified in the SAP.
Measure: Geometric Mean (95% Confidence Interval); unit: Units/milliliter (U/mL)
Arm/Group | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo
Number analyzed (Participants) | 91 | 92
Units/milliliter (U/mL)
  At Birth | 5576.4 [4246.2 to 7323.2] | 19.4 [10.2 to 37.0]
  6 months of age: number analyzed (Participants) | 83 | 69
  6 months of age | 311.1 [235.8 to 410.5] | 22.0 [11.4 to 42.7]

21. Secondary Outcome: GMFR of Full-Length S-Binding IgG Levels From Birth to 6 Months of Age in Infant Participants Born to Evaluable Maternal Participants
Description: GMFRs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. GMFR of full-length S-binding IgG levels from birth to 6 months of age in infant participants born to evaluable maternal participants was reported in this outcome measure.
Time Frame: From birth to 6 months of age
Population: All infant participants born to evaluable immunogenicity maternal participants and had no important protocol deviations as determined by the clinician. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. HIV positive participants were excluded from analysis as pre-specified in the SAP.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo
Number analyzed (Participants) | 75 | 65
Fold rise | 0.1 [0.0 to 0.1] | 0.6 [0.3 to 1.3]

ADVERSE EVENTS:
Time Frame: Maternal participants-Local reactions/systemic events: From Day (D) 1 to 7 after dose 1 and 2; SAEs: from dose 1 on D 1 up to 6 months (M) after delivery (approx 10 M) (BNT162b2 30 mcg) and up to 1 M after delivery (approx 5 M) (placebo); placebo then BNT162b2: from Dose 3 up to 1 M after Dose 4 (approx 2 M); other AEs: from dose 1 up to 1 M after dose 2 (approx 2 M); (placebo then BNT162b2): from Dose 3 up to 1 M after Dose 4 (approx 2 M). For infants-SAEs and AESIs: from birth up to 6 M of age
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other, or a participant may have experienced both serious and non-serious event. Safety population for maternal and infants was evaluated. Systematic events include local reactions and systemic events recorded by participants in e-diary and non-systematic events include all other AEs.
Groups:
- Maternal Participants: BNT162b2 30 mcg (Blinded Phase): Maternal participants received two doses of BNT162b2 30 micrograms (mcg) as an intramuscular injection separated by 21 days during their 24 to 34 weeks gestation in the blinded phase. Participants were followed-up until 6 months post-delivery. HIV positive maternal participants were excluded.
- Maternal Participants: Placebo (Blinded Phase): Maternal participants received two doses of placebo as an intramuscular injection separated by 21 days during their 24 to 34 weeks gestation in the blinded phase. HIV positive maternal participants were excluded.
- Maternal Participants: Placebo Then BNT162b2 (Unblinded Phase): Participants who originally received 2 doses of blinded placebo were administered 2 doses of 30 mcg BNT162b2 vaccine as intramuscular injection separated by 21 days after unblinding at 1 month post-delivery. Participants were followed-up until 1 month after last vaccination. HIV positive maternal participants were excluded.
- Infant Participants: BNT162b2 30 mcg: Infant participants who were born to maternal participants vaccinated with BNT162b2 30 mcg during pregnancy were included. Infant participants were followed up to 6 months of age. HIV positive infant participants born to HIV positive maternal participants were excluded.
- Infant Participants: Placebo: Infant participants who were born to maternal participants vaccinated with placebo during pregnancy were included. Infant participants were followed up to 6 months of age. HIV positive infant participants born to HIV positive maternal participants were excluded.
- HIV Positive Maternal Participants: BNT162b2 30 mcg (Blinded Phase): Maternal participants who were HIV positive received two doses of BNT162b2 30 micrograms (mcg) as an intramuscular injection separated by 21 days during their 24 to 34 weeks gestation in the blinded phase. Participants were followed-up until 6 months post-delivery.
- HIV Positive Maternal Participants: Placebo (Blinded Phase): Maternal participants who were HIV positive received two doses of placebo as an intramuscular injection separated by 21 days during their 24 to 34 weeks gestation in the blinded phase.
- HIV Positive Maternal Participants: Placebo Then BNT162b2 (Unblinded Phase): HIV positive maternal participants who originally received 2 doses of blinded placebo were administered 2 doses of 30 mcg BNT162b2 vaccine as intramuscular injection separated by 21 days after unblinding at 1 month post-delivery. Participants were followed-up until 1 month after last vaccination.
- HIV Positive Infant Participants: BNT162b2 30 mcg: Infant participants who were born to HIV positive maternal participants vaccinated with BNT162b2 30 mcg during pregnancy were included. Infant participants were followed up to 6 months of age.
- HIV Positive Infant Participants: Placebo: Infant participants who were born to HIV positive maternal participants vaccinated with placebo during pregnancy were included. Infant participants were followed up to 6 months of age.
Arm/Group | Maternal Participants: BNT162b2 30 mcg (Blinded Phase) | Maternal Participants: Placebo (Blinded Phase) | Maternal Participants: Placebo Then BNT162b2 (Unblinded Phase) | Infant Participants: BNT162b2 30 mcg | Infant Participants: Placebo | HIV Positive Maternal Participants: BNT162b2 30 mcg (Blinded Phase) | HIV Positive Maternal Participants: Placebo (Blinded Phase) | HIV Positive Maternal Participants: Placebo Then BNT162b2 (Unblinded Phase) | HIV Positive Infant Participants: BNT162b2 30 mcg | HIV Positive Infant Participants: Placebo
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/163 | 0/144 | 0/156 | 1/159 | 0/12 | 0/10 | 0/8 | 1/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 21/161 | 23/163 | 0/144 | 21/156 | 24/159 | 2/12 | 4/10 | 0/8 | 1/11 | 2/9
Other Adverse Events (participants affected / at risk) | 143/161 | 119/163 | 21/144 | 29/156 | 33/159 | 12/12 | 10/10 | 1/8 | 1/11 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maternal Participants: BNT162b2 30 mcg (Blinded Phase) (N=161) | Maternal Participants: Placebo (Blinded Phase) (N=163) | Maternal Participants: Placebo Then BNT162b2 (Unblinded Phase) (N=144) | Infant Participants: BNT162b2 30 mcg (N=156) | Infant Participants: Placebo (N=159) | HIV Positive Maternal Participants: BNT162b2 30 mcg (Blinded Phase) (N=12) | HIV Positive Maternal Participants: Placebo (Blinded Phase) (N=10) | HIV Positive Maternal Participants: Placebo Then BNT162b2 (Unblinded Phase) (N=8) | HIV Positive Infant Participants: BNT162b2 30 mcg (N=11) | HIV Positive Infant Participants: Placebo (N=9)
Bradycardia fetal (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non reassuring fetal heart rate pattern (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergic gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meconium plug syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endometritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Neonatal pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Injury to brachial plexus due to birth trauma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Traumatic intracranial hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fetal heart rate abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ultrasound fetal abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrested labor (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Failed induction of labor (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meconium stain (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Omphalorrhexis (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 7 | 4 | 0 | 0 | 0 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine disorder (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoperfusion (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subgaleal hemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Congenital rubella syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DiGeorge's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Microcephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucopolysaccharidosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syndactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycemia neonatal (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy neonatal (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxic-ischemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failed trial of labor (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maternal Participants: BNT162b2 30 mcg (Blinded Phase) (N=161) | Maternal Participants: Placebo (Blinded Phase) (N=163) | Maternal Participants: Placebo Then BNT162b2 (Unblinded Phase) (N=144) | Infant Participants: BNT162b2 30 mcg (N=156) | Infant Participants: Placebo (N=159) | HIV Positive Maternal Participants: BNT162b2 30 mcg (Blinded Phase) (N=12) | HIV Positive Maternal Participants: Placebo (Blinded Phase) (N=10) | HIV Positive Maternal Participants: Placebo Then BNT162b2 (Unblinded Phase) (N=8) | HIV Positive Infant Participants: BNT162b2 30 mcg (N=11) | HIV Positive Infant Participants: Placebo (N=9)
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (DIARRHEA) (Gastrointestinal disorders) | 24 | 21 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (VOMITING) (Gastrointestinal disorders) | 18 | 16 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Chills (CHILLS) (General disorders) | 28 | 10 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Erythema (REDNESS) (General disorders) | 11 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (FATIGUE) (General disorders) | 101 | 82 | 0 | 0 | 0 | 8 | 8 | 0 | 0 | 0
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 138 | 30 | 13 | 0 | 0 | 12 | 4 | 0 | 0 | 0
Pyrexia (FEVER) (General disorders) | 6 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling (SWELLING) (General disorders) | 17 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcus test positive (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (NEW OR WORSENED JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 22 | 13 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (NEW OR WORSENED MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 53 | 26 | 0 | 0 | 0 | 5 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 7 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (HEADACHE) (Nervous system disorders) | 85 | 72 | 0 | 0 | 0 | 7 | 7 | 0 | 0 | 0
Abnormal labor (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Episiotomy (Surgical and medical procedures) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Congenital naevus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinemia neonatal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0
Apgar score low (Investigations) | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Hypoglycemia neonatal (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 12 | 13 | 0 | 0 | 0 | 0 | 1
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 1 | 0
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor (or its agents) has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04754594/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT04754594/SAP_001.pdf